CLINICAL TRIAL: NCT02812160
Title: A Randomized, Controlled, Multicenter Study Comparing the Spatz3 Adjustable Balloon System Plus Diet and Exercise to Diet and Exercise Alone
Brief Title: Spatz Adjustable Balloon for Obesity (SABO)
Acronym: SABO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spatz FGIA, Inc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Spatz-160061
Record Dates: First submitted 2016-05-25; First posted 2016-06-24 (Estimated); Results first posted 2021-05-28 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Obesity
Keywords: weight loss
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Spatz3 Adjustable Balloon (Active Comparator): Spatz3 Adjustable Balloon with Dietary and exercise counselling
  Interventions: Device: Spatz3 Adjustable Balloon
- Control (No Intervention): Dietary and Exercise counselling

INTERVENTIONS:
Device: Spatz3 Adjustable Balloon — An adjustable intragastric balloon for weight loss that can have the balloon volume increased or decrease as needed
  Arms: Spatz3 Adjustable Balloon

SUMMARY:
The purpose of this study is to determine whether the Spatz3 Adjustable balloon, a non-surgical device, is effective in the treatment of obesity.

DETAILED DESCRIPTION:
Device Name: Spatz3 Adjustable Balloon System® (Spatz3) Clinical Phase: Pivotal Trial Design: Multicenter open-label randomized controlled trial Trial Participants: Adults, ages 22-65, with a BMI ≥ 30 and < 40 who have failed to achieve and maintain weight-loss with a weight control program Control group: Supervised diet and exercise Planned sample size: 282 subjects randomized 2:1 to device/control study treatment duration: 32 weeks Primary endpoint: Percent change in total body weight (%TBL) at 32 weeks

ELIGIBILITY:
Inclusion Criteria:

1. Age 22 - 65
2. BMI ≥ 30 and <40
3. Willingness to comply with the substantial lifelong dietary restrictions required by the procedure
4. History of obesity (BMI ≥ 30) for at least 2 years
5. History of failure with non-surgical weight loss methods
6. Willingness to follow protocol requirements, including signed informed consent, routine follow-up schedule, completing laboratory tests, completing diet counseling
7. Residing within a reasonable distance from the investigator's office and able to travel to the investigator to complete all routine follow- up visits
8. Ability to give informed consent
9. Women of childbearing potential (i.e., not post-menopausal or surgically sterilized) must agree to use adequate birth control methods. Acceptable birth control methods are limited to hormonal contraceptives (oral, flexible vaginal ring, skin patch, injection), diaphragms, IUDs, condoms with or without spermicide, and voluntary abstinence. The method of birth control must be documented and verified at follow-up. Should a treatment arm subject become pregnant during the implantation period, the balloon will be extracted during the second trimester - the timing of which will be determined via consultation with the subject's obstetrician.

Exclusion Criteria:

1. Prior gastrointestinal surgery with sequelae, i.e. obstruction, and/or adhesive peritonitis or known abdominal adhesions.
2. Prior open or laparoscopic bariatric surgery.
3. Prior surgery of any kind on the esophagus, stomach or any type of hiatal hernia surgery.
4. Any inflammatory disease of the gastrointestinal tract including esophagitis, Barrett's esophagus, gastric ulceration, duodenal ulceration, cancer or specific inflammation such as Crohn's disease.
5. Potential upper gastrointestinal bleeding conditions such as esophageal or gastric varices, congenital or acquired intestinal telangiectasis, or other congenital anomalies of the gastrointestinal tract such as atresias or stenoses.
6. A gastric mass.
7. A hiatal hernia > 2cm or severe or intractable gastro-esophageal reflux symptoms.
8. Acid reflux symptoms to any degree that require more than one medication for symptom control.
9. A structural abnormality in the esophagus or pharynx such as a stricture or diverticulum that could impede passage of the balloon alongside the endoscope.
10. Achalasia or any other severe esophageal motility disorder that may pose a safety risk during the removal of the device
11. Severe coagulopathy.
12. Insulin-dependent diabetes (either Type 1 or Type 2) or a significant likelihood of requiring insulin treatment in the following 12 months.
13. Subjects with any serious health condition unrelated to their weight that would increase the risk of endoscopy
14. Chronic abdominal pain
15. Motility disorders of the GI tract such as gross esophageal motility disorders, gastroparesis or intractable constipation
16. Hepatic insufficiency or cirrhosis
17. Serious or uncontrolled psychiatric illness or disorder that could compromise patient understanding of or compliance with follow up visits and removal of the device after 8 months.
18. Alcoholism or drug addiction.
19. Patients unwilling to participate in an established medically-supervised diet and behavior modification program, with routine medical follow-up.
20. Patients receiving daily prescribed treatment with aspirin, anti-inflammatory agents, anticoagulants or other gastric irritants.
21. Patients who are unable or unwilling to take prescribed proton pump inhibitor medication for the duration of the device implant.
22. Patients who are known to have, or suspected to have, an allergic reaction to materials contained in the system.
23. Patients who have ever developed a serotonin syndrome and are currently taking any drug known to affect the levels of serotonin in the body [e.g., selective serotonin reuptake inhibitors (SSRIs), serotonin-norepinephrine reuptake inhibitors (SNRIs), monoamine oxidase inhibitors (MAOIs)] should not undergo placement of the device.
24. Patients who are pregnant or breast-feeding.
25. Subjects with Severe cardiopulmonary disease or other serious organic disease which might include known history of coronary artery disease, Myocardial infarction within the past 6 months, poorly-controlled hypertension, required use of NSAIDs
26. Subjects who have tested positive for H. Pylori.
27. Subjects taking medications on specified hourly intervals that may be affected by changes to gastric emptying, such as anti-seizure or anti-arrhythmic medications
28. Subjects who are taking corticosteroids, immunosuppressants, and narcotics
29. Subjects who are taking diet pills
30. Use of an intragastric device prior to this study due to the potential increase in risk associated with implantation of a balloon in a previously instrumented and possibly scarred stomach.
31. Participation in any clinical study which could affect weight loss within the past 6 months due to the potential to confound findings.
32. Symptomatic congestive heart failure, cardiac arrhythmia or unstable coronary artery disease.
33. Pre-existing respiratory disease such as chronic obstructive pulmonary disease (COPD), pneumonia or cancer.
34. Diagnosis of autoimmune connective tissue disorder (e.g. lupus, erythematous, scleroderma) or immunocompromised.
35. Life expectancy less than 1 year or severe renal, hepatic, pulmonary or other medical condition, in the opinion of the investigator because of an increased risk profile.
36. Specific diagnosed genetic or hormonal cause for obesity such as hypothyroidism or Prader Willi syndrome
37. Eating disorders including night eating syndrome (NES), bulimia, binge eating disorder, or compulsive overeating
38. Known history of endocrine disorders affecting weight

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2016-09-12 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barham AbuDayyeh, MD, Principal Investigator — Mayo Clinic; Christopher C Thompson, MD, Principal Investigator — Brigham and Women's Hospital
Locations (7):
- United States (7):
  - University of Chicago, Chicago, Illinois
  - Surgical Specialists of Louisiana, Metairie, Louisiana
  - Endoscopic MicroSurgery Associates, Towson, Maryland
  - Brigham and Womans Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - NY Manhattan VA Hospital, New York, New York
  - Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Abu Dayyeh BK, Maselli DB, Rapaka B, Lavin T, Noar M, Hussan H, Chapman CG, Popov V, Jirapinyo P, Acosta A, Vargas EJ, Storm AC, Bazerbachi F, Ryou M, French M, Noria S, Molina D, Thompson CC. Adjustable intragastric balloon for treatment of obesity: a multicentre, open-label, randomised clinical trial. Lancet. 2021 Nov 27;398(10315):1965-1973. doi: 10.1016/S0140-6736(21)02394-1. Epub 2021 Nov 15. PMID 34793746

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Spatz3 Adjustable Balloon | Control
Started | 187 | 101
Completed | 187 | 101
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The overall number of baseline participants does not differ from the number of participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Spatz3 Adjustable Balloon | Control | Total
Number analyzed (Participants) | 187 | 101 | 288
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 187 | 101 | 288
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (8.9) | 44.0 (8.9) | 44.3 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 162 | 90 | 252
  Male | 25 | 11 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 49 | 26 | 75
  White | 132 | 72 | 204
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 2 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 187 | 101 | 288
BMI [Mean (Standard Deviation); unit: Kg/m^2] — Body Mass Index BMI = kg/m2 where kg is a person's weight in kilograms and m2 is their height in metres
  Kg/m^2 | 35.8 (2.6) | 35.8 (2.7) | 35.8 (2.6)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Total Body Weight (%TBL) .
Description: The mean %TBL in the Spatz3 group should exceed the %TBL control group by 4.5%.
Time Frame: 32 weeks
Measure: Mean (Standard Deviation); unit: TBL%
Arm/Group | Spatz3 Adjustable Balloon | Control
Number analyzed (Participants) | 187 | 101
TBL% | 15.0 (7.2) | 3.3 (5.6)

ADVERSE EVENTS:
Time Frame: 32 weeks
Arm/Group | Spatz3 Adjustable Balloon | Control
All-Cause Mortality (participants affected / at risk) | 0/187 | 0/101
Serious Adverse Events (participants affected / at risk) | 10/187 | 1/101
Other Adverse Events (participants affected / at risk) | 184/187 | 32/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Spatz3 Adjustable Balloon (N=187) | Control (N=101)
Gastrointestinal disorders (Gastrointestinal disorders) | 7 (24) | 1 (1) — Nausea, Vomiting, Abdominal pain, Diarrhoea, Abdominal discomfort, Gastrooesophageal reflux , disease, Abdominal pain upper, Colitis
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 4 (5) | 0 (0) — Dehydration, Failure to thrive, Hypokalaemia
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Spatz3 Adjustable Balloon (N=187) | Control (N=101)
Gastrointestinal disorders (Gastrointestinal disorders) | 184 (2522) | 32 (84)

LIMITATIONS AND CAVEATS:
There are no overall Limitations and Caveats

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-11): https://cdn.clinicaltrials.gov/large-docs/60/NCT02812160/Prot_SAP_000.pdf